CLINICAL TRIAL: NCT07029451
Title: Prospective, Post-authorisation, Multi-centre, Non-interventional Study to Investigate REKOVELLE in Chinese Women Undergoing Assisted Reproductive Technologies: Effectiveness, Safety, and Patterns of Use in Real-world Practice
Brief Title: To Investigate REKOVELLE in Chinese Women Undergoing Assisted Reproductive Technologies: Effectiveness, Safety, and Patterns of Use in Real-world Practice
Acronym: LYCHEE
Status: Recruiting | Type: Observational
Sponsor: Ferring Pharmaceuticals (Industry)
Responsible Party: Sponsor
Other Study IDs: 000442
Record Dates: First submitted 2025-06-10; First posted 2025-06-19 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Infertility
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a multi-centre prospective non-interventional trial to assess the pattern of use of REKOVELLE® in Women Undergoing In Vitro Fertilisation (IVF) or Intracytoplasmic Sperm Injection (ICSI) Procedures in Routine Clinical Practice.

There will be approximately 2500 patients initiated with REKOVELLE® treatment and enrolled in 30-50 sites in China. The total duration of the study will be approximately 35 months.

ELIGIBILITY:
Inclusion Criteria:

* Women who meet all the following criteria are eligible for participation:

  * At least 20 years of age (including the 20th birthday) when signing informed consent
  * Prescribed REKOVELLE for the first time in controlled ovarian stimulation for in vitro fertilisation (IVF) or intracytoplasmic sperm injection (ICSI) cycles
  * Willing and able to provide written informed consent

Exclusion Criteria:

* Women who meet any of the following criteria are not eligible for participation:

  * Previously undergone more than 1 controlled ovarian stimulation cycles for IVF or ICSI
  * Currently participating in an interventional clinical study for which treatment with medication is mandated
  * Currently undergoing ovarian stimulation for fertility preservation or oocytes donation
  * Contraindications for the use of REKOVELLE

Min Age: 20 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: Women eligible for enrolment in the study are those scheduled for their first REKOVELLE treatment, with no more than one prior COS cycle for IVF or ICSI, and who meet the inclusion and exclusion criteria. Data from approximately 2,500 patients will be collected.
Sampling Method: Non-Probability Sample
Enrollment: 2500 (Estimated)
Dates: Start 2025-08-05 (Actual); Primary Completion 2028-09-30 (Estimated); Study Completion 2028-09-30 (Estimated)

PRIMARY OUTCOMES:
Live Birth Rate per initiated stimulation cycles | Up to 15 months

SECONDARY OUTCOMES:
Serum oestradiol levels | Up to 20 days
  Serum oestradiol levels on days of stimulation initiation (before treatment) and at end-of-stimulation
Progesterone (P4) levels | Up to 20 days
  Progesterone (P4) levels on days of stimulation initiation (before treatment) and at end-of-stimulation
Cycle cancellation rate and reasons for cycle cancellation | Up to 28 days
Number of oocytes retrieved | Up to 22 days
Number of metaphase II (MII) oocytes | Up to 22 days
  Number of metaphase II (MII) oocytes for intracytoplasmic sperm injection (ICSI)
Number of embryos on Day 3 after oocyte retrieval | Day 3 after oocyte retrieval
Number of embryos on Day 5 after oocyte retrieval | Day 5 after oocyte retrieval
Number of transferred embryos | Up to 28 days
Number of transferred blastocysts | Up to 28 days
Transfer cancellation rate and reasons for transfer cancellation | Up to 28 days
Implantation rate | Up to 28 days
  Number of gestational sacs, embryos or blastocysts transferred
Positive beta-human chorionic gonadotropin (βhCG) test rate | 11-15 days after transfer
Clinical pregnancy rate | 4 to 6 weeks after transfer
  At least one intrauterine gestational sac 4-6 weeks after transfer
Vital pregnancy rate | 4 to 6 weeks after transfer
  At least 1 intrauterine gestational sac with fetal heartbeat 4-6 weeks after transfer
Ongoing pregnancy rate | 9 to 11 weeks after transfer
  At least 1 intrauterine viable fetus 9-11 weeks after transfer
Cumulative ongoing pregnancy rate | 9 to 11 days
Time to pregnancy | 4 to 6 weeks after transfer
  Time to pregnancy from stimulation initiation to ongoing pregnancy
Pregnancy loss rate | Up to 10 - 11 weeks after transfer
Live birth rate per initiated stimulation cycles with fresh transfer cycles | More than 20 weeks after transfer
Cumulative live birth rate per initiated stimulation cycles | More than 20 weeks after transfer
Frequency and severity of adverse drug reactions | During 1st cycle with REKOVELLE (each cycle range is 5-20 days, average 9 days), Up to 10-11 weeks after transfer
Frequency of preventive interventions for early ovarian hyperstimulation syndrome (OHSS) | During 1st cycle with REKOVELLE (each cycle range is 5-20 days, average 9 days), Up to 10-11 weeks after transfer
Frequency of early OHSS | Up to 9 days after triggering of final follicular maturation
Frequency of late OHSS | Up to 10-11 weeks after transfer
Use of luteinising hormone (LH) surge suppression protocols | Up to 22 days
Daily dose of REKOVELLE | Up to 22 days
  Use of REKOVELLE protocol, including daily dose
Total dose of REKOVELLE | Up to 22 days
  Use of REKOVELLE protocol including total dose
Stimulation duration | Up to 22 days
  Stimulation duration following use of REKOVELLE protocol
Use of any other concomitant ovarian stimulation agent, including daily dose, total dose, and stimulation duration | Up to 22 days
Use of follicle maturation triggering protocol | Up to 22 days

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Compliance, Study Director — Ferring Pharmaceuticals
Locations (28):
- China (28):
  - The First Affiliated Hospital of Anhui Medical University, Hefei, Anhui
  - Maanshan Maternal and Child Health Care Hospital, Ma’anshan, Anhui
  - Beijing Obstetrics And Gynecology Hospital Capital Medical University, Beijing, Beijing Municipality
  - Beijing Chaoyang Hospital (Beijing), Chaoyang, Beijing Municipality
  - Peking University First Hospital, Xicheng, Beijing Municipality
  - 6th Affiliated Hospital of Sun Yat Sen University, Guangzhou, Guandong
  - 3rd Affiliated Hospital of Guangzhou Medical University (Guangzhou), Guangzhou, Guangdong
  - The First Affiliated Hospital of Shantou University Medical College, Shantou, Guangdong
  - The Second Nanning People's Hospital, Nanning, Guangxi
  - Tongji Hospital Tongji Medical College of Hust, Wuhan, Hubei
  - Hubei Maternal and Child Health Hospital, Wuhan, Hubei
  - Reproductive & Genetic hospital Of CITIC-Xiangya, Changsha, Hunan
  - 1st Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - General Hospital of Ningxia Medical University, Yinchuan, Ningxia
  - The Second Affiliated Hospital of Air Force Medical University, Xi'an, Shaanxi
  - Binzhou Medical University Hospital, Binzhou, Shandong
  - Reproductive Hospital Affiliated to Shandong University, Jinan, Shandong
  - Affiliated Hospital of Jining Medical University, Jining, Shandong
  - Shanghai First Maternal and Child Health Hospital, Shanghai, Shanghai Municipality
  - Northwest Women's and Children's Hospital, Xi’an, Shanxi
  - Tianjin Medical University General Hospital (Heping District), Xiaobailou, Tianjin Municipality
  - Women's hospital School of Medicine Zhejiang University, Hangzhou, Zhejiang
  - Peking University Third Hospital (Beijing), Beijing
  - Zhejiang Provincial People's Hospital, Hangzhou
  - Jinhua People's Hospital, Jinhua
  - The Peoples Hospital of Guangxi Zhuang Autonomous Region, Nanning
  - The Reproduction Hospital of Guangxi Zhuang Autonomous Region, Nanning
  - Zhongshan Hospital Affiliated to Fudan University, Shanghai

IPD SHARING:
Plan to Share IPD: No